CLINICAL TRIAL: NCT01354496
Title: LY2409021 Formulation Bridging and Food Effect Study
Brief Title: A Study of LY2409021 Formulations and the Effect of Food
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 14194; I1R-FW-GLBQ (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-05-13; First posted 2011-05-17 (Estimated); Results first posted 2019-03-11 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2018-11

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers; Bioavailability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1 - LY2409021 reference form (Experimental): A 20 milligram (mg) LY2409021 dose, reference form administered orally in the fasted state
  Interventions: Drug: LY2409021 Reference Form
- Cohort 1 - LY2409021 medium test form fed (Experimental): Single 20 mg LY2409021 test form with medium particle size administered orally immediately after ingestion of a standardized high-fat meal
  Interventions: Drug: LY2409021 Test-Med Formulation (medium particle size)
- Cohort 1 - LY2409021 medium test form fasted (Experimental): Single 20 mg LY2409021 test form with medium particle size administered orally in the fasted state
  Interventions: Drug: LY2409021 Test-Med Formulation (medium particle size)
- Cohort 2 - LY2409021 low test form fasted (Experimental): Single 20 mg LY2409021 test form with low particle size administered orally in the fasted state
  Interventions: Drug: LY2409021 Test-Low Formulation (low particle size)
- Cohort 2 - LY2409021 medium test form fasted (Experimental): Single 20 mg LY2409021 test form with medium particle size administered orally in the fasted state
  Interventions: Drug: LY2409021 Test-Med Formulation (medium particle size)
- Cohort 2 - LY2409021 high test form fasted (Experimental): Single 20 mg LY2409021 test form with high particle size administered orally in the fasted state
  Interventions: Drug: LY2409021 Test-High Formulation (high particle size)

INTERVENTIONS:
Drug: LY2409021 Reference Form — Administered orally
  Arms: Cohort 1 - LY2409021 reference form
Drug: LY2409021 Test-Med Formulation (medium particle size) — Administered orally
  Arms: Cohort 1 - LY2409021 medium test form fasted; Cohort 1 - LY2409021 medium test form fed; Cohort 2 - LY2409021 medium test form fasted
Drug: LY2409021 Test-High Formulation (high particle size) — Administered orally
  Arms: Cohort 2 - LY2409021 high test form fasted
Drug: LY2409021 Test-Low Formulation (low particle size) — Administered orally
  Arms: Cohort 2 - LY2409021 low test form fasted

SUMMARY:
The purposes of this study are to compare how much of LY2409021 enters the bloodstream and how long the body takes to get rid of the drug when different formulations of LY2409021 are given, and when LY2409021 is taken with or without food.

The study will be conducted in 2 cohorts. Each cohort will have 3 study periods consisting of 3 formulations of LY2409021. Participants in each cohort will receive the same all 3 formulations using a randomized sequence crossover design. There is a washout period of at least 14 days between dosing periods.

There will be an interim analysis after Cohort 1 completes study Period 2. Cohort 2 will not begin enrolling until this analysis is complete. The need to enroll Cohort 2 will be determined by the outcome of the interim analysis.

ELIGIBILITY:
Inclusion Criteria:

* Must be healthy male or a healthy female who cannot become pregnant
* Must have body mass index (BMI) of 18.5 to 32 kilograms per meter squared (kg/m²), inclusive
* Blood pressure as well as blood and urine laboratory test results must be acceptable for the study
* The veins must be suitable for easy blood collection
* Must be willing to be available for the whole study and be willing to follow study procedures

Exclusion Criteria:

* Were in another new drug or medical research study in the last 30 days
* Have previously taken part in this study or any other study with LY2409021
* Have taken LY2409021, or drugs similar to LY2409021 before and was found to be allergic to the drug
* Currently have or used to have health problems or laboratory test results that in the opinion of the doctor, could interfere with understanding the results of this study
* Electrocardiogram (ECG) readings are not suitable for the study
* Are infected with hepatitis B
* Are infected with human immunodeficiency disease virus (HIV)
* Are using or intend to use over-the-counter medication or prescription medications within 14 days, from the start of the first study dosing until end of study
* Have a regular alcohol intake greater than 21 units per week (males) and 14 units per week (females) or are not willing to abstain from alcohol while in the research unit
* Smoke more than 10 cigarettes per day or are not willing to abstain from smoking while at the clinic
* Have a history of drug or alcohol abuse
* Have donated 450 milliliters (mL) or more of blood in the last 3 months
* Are unwilling or unable to comply with dietary requirements/restrictions during the study
* The study doctor thinks the participant should not participate for any other reasons

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your person physician., Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- LY2409021 Cohort 1: Sequence 1: Sequence 1: (Period 1:reference capsules fasting, then Period 2: test-medium tablet fasting, then Period 3: test-medium tablet after high-fat meal).
  There was a washout period of at least 14 days between interventions. Description of interventions: reference capsules fasting [20-milligram (mg) LY2409021 dose, administered orally, once in fasted state], test-medium tablet fasting (20-mg LY2409021 tablet, medium particle size, administered orally, once in fasted state), and test-medium tablet after high-fat meal (20-mg LY2409021 tablet, medium particle size, administered orally, once, immediately after standardized high-fat meal).
- LY2409021 Cohort 1: Sequence 2: Sequence 2: (Period 1: test-medium tablet fasting, then Period 2: test-medium tablet after high-fat meal, then Period 3: reference capsules fasting).
  There was a washout period of at least 14 days between interventions. Description of interventions: reference capsules fasting [20-milligram (mg) LY2409021 dose, administered orally, once in fasted state], test-medium tablet fasting (20-mg LY2409021 tablet, medium particle size, administered orally, once in fasted state), and test-medium tablet after high-fat meal (20-mg LY2409021 tablet, medium particle size, administered orally, once, immediately after standardized high-fat meal).
- LY2409021 Cohort 1: Sequence 3: Sequence 3: (Period 1:test-medium tablet after high-fat meal, then Period 2: reference capsules fasting, then Period 3: test-medium tablet fasting).
  There was a washout period of at least 14 days between interventions. Description of interventions: reference capsules fasting [20-milligram (mg) LY2409021 dose, administered orally, once in fasted state], test-medium tablet fasting (20-mg LY2409021 tablet, medium particle size, administered orally, once in fasted state), and test-medium tablet after high-fat meal (20-mg LY2409021 tablet, medium particle size, administered orally, once, immediately after standardized high-fat meal).
- LY2409021 Cohort 2: Sequence 4: Sequence 4: (Period 1: test-medium tablet fasting then, Period 2: test-high tablet fasting, then Period 3: test-low tablet fasting) There was a washout period of at least 14 days between interventions. Description of interventions: test-low tablet fasting (single 20-mg LY2409021 tablet of a low particle size, administered orally in a fasted state), test-medium tablet fasting (single 20-mg LY2409021 tablet of a medium particle size, administered orally, once in a fasted state), and test-high tablet fasting (single 20-mg LY2409021 tablet of a high particle size administered orally, once in a fasted state).
- LY2409021 Cohort 2: Sequence 5: Sequence 5: (Period 1: test-high tablet fasting then, Period 2: test-low tablet fasting, then Period 3: test-medium tablet fasting) There was a washout period of at least 14 days between interventions. Description of interventions: test-low tablet fasting (single 20-mg LY2409021 tablet of a low particle size, administered orally in a fasted state), test-medium tablet fasting (single 20-mg LY2409021 tablet of a medium particle size, administered orally, once in a fasted state), and test-high tablet fasting (single 20-mg LY2409021 tablet of a high particle size administered orally, once in a fasted state).
- LY2409021 Cohort 2: Sequence 6: Sequence 6: (Period1: test-low tablet fasting, then Period 2: test-medium tablet fasting, then Period 3: test-high tablet fasting).
  There was a washout period of at least 14 days between interventions. Description of interventions: test-low tablet fasting (single 20-mg LY2409021 tablet of a low particle size, administered orally in a fasted state), test-medium tablet fasting (single 20-mg LY2409021 tablet of a medium particle size, administered orally, once in a fasted state), and test-high tablet fasting (single 20-mg LY2409021 tablet of a high particle size administered orally, once in a fasted state).
Period: Period 1
Arm/Group | LY2409021 Cohort 1: Sequence 1 | LY2409021 Cohort 1: Sequence 2 | LY2409021 Cohort 1: Sequence 3 | LY2409021 Cohort 2: Sequence 4 | LY2409021 Cohort 2: Sequence 5 | LY2409021 Cohort 2: Sequence 6
Started | 6 | 6 | 6 | 6 | 5 | 6
Received at Least 1 Dose of Study Drug | 6 | 6 | 6 | 6 | 5 | 6
Completed | 6 | 6 | 4 | 6 | 5 | 6
Not Completed | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0
Period: Washout (at Least 14 Days)
Arm/Group | LY2409021 Cohort 1: Sequence 1 | LY2409021 Cohort 1: Sequence 2 | LY2409021 Cohort 1: Sequence 3 | LY2409021 Cohort 2: Sequence 4 | LY2409021 Cohort 2: Sequence 5 | LY2409021 Cohort 2: Sequence 6
Started | 6 | 6 | 4 | 6 | 5 | 6
Completed | 6 | 6 | 4 | 6 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | LY2409021 Cohort 1: Sequence 1 | LY2409021 Cohort 1: Sequence 2 | LY2409021 Cohort 1: Sequence 3 | LY2409021 Cohort 2: Sequence 4 | LY2409021 Cohort 2: Sequence 5 | LY2409021 Cohort 2: Sequence 6
Started | 6 | 6 | 4 | 6 | 5 | 6
Completed | 6 | 6 | 4 | 5 | 5 | 6
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Period: Washout (at Least 14 Days)
Arm/Group | LY2409021 Cohort 1: Sequence 1 | LY2409021 Cohort 1: Sequence 2 | LY2409021 Cohort 1: Sequence 3 | LY2409021 Cohort 2: Sequence 4 | LY2409021 Cohort 2: Sequence 5 | LY2409021 Cohort 2: Sequence 6
Started | 6 | 6 | 4 | 5 | 5 | 6
Completed | 6 | 5 | 4 | 4 | 5 | 6
Not Completed | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Scheduling Conflict | 0 | 1 | 0 | 1 | 0 | 0
Period: Period 3
Arm/Group | LY2409021 Cohort 1: Sequence 1 | LY2409021 Cohort 1: Sequence 2 | LY2409021 Cohort 1: Sequence 3 | LY2409021 Cohort 2: Sequence 4 | LY2409021 Cohort 2: Sequence 5 | LY2409021 Cohort 2: Sequence 6
Started | 6 | 5 | 4 | 4 | 5 | 6
Completed | 6 | 5 | 4 | 4 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized participants who received at least 1 dose of study drug.
Groups:
- LY2409021 Cohort 1: Participants randomized to 1 of 3 sequences and received a single but different intervention per period: Sequence 1 (reference capsules fasting, then test-medium tablet fasting, then test-medium tablet after high-fat meal), Sequence 2 (test-medium tablet fasting, then test-medium tablet after high-fat meal, then reference capsules fasting), or Sequence 3 (test-medium tablet after high-fat meal, then reference capsules fasting, then test-medium tablet fasting).
  There was a washout period of at least 14 days between interventions. Description of interventions: reference capsules fasting [20-milligram (mg) LY2409021 dose, administered orally, once in fasted state], test-medium tablet fasting (20-mg LY2409021 tablet, medium particle size, administered orally, once in fasted state), and test-medium tablet after high-fat meal (20-mg LY2409021 tablet, medium particle size, administered orally, once, immediately after standardized high-fat meal).
- LY2409021 Cohort 2: Participants randomized to 1 of 3 sequences and received a single but different intervention per period: Sequence 4 (test-medium tablet fasting then, test-high tablet fasting, then test-low tablet fasting), Sequence 5 (test-high tablet fasting then, test-low tablet fasting, then test-medium tablet fasting), or Sequence 6 (test-low tablet fasting, then test-medium tablet fasting, then test-high tablet fasting).
  There was a washout period of at least 14 days between interventions. Description of interventions: test-low tablet fasting (single 20-mg LY2409021 tablet of a low particle size, administered orally in a fasted state), test-medium tablet fasting (single 20-mg LY2409021 tablet of a medium particle size, administered orally, once in a fasted state), and test-high tablet fasting (single 20-mg LY2409021 tablet of a high particle size administered orally, once in a fasted state).
- Total: Total of all reporting groups
Arm/Group | LY2409021 Cohort 1 | LY2409021 Cohort 2 | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.4 (10.7) | 32.6 (9.7) | 33.6 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 18 | 15 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 18 | 17 | 35
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 18 | 17 | 35

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics, Area Under the Concentration-Time Curve (AUC): Medium Test Form to Reference Form
Description: AUC from time 0 to infinity (AUC0-∞).
Time Frame: Periods 1, 2, 3 (predose, 0.5, 1, 2, 4, 6, 8, 10, 12, 18, 24, 36, 48, 72, 96, 144, 192, 240, 288, and 336 hours postdose)
Population: Randomized participants in Cohort 1 who received the specified study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*hr/mL)
Groups:
- LY2409021 Cohort 1 (Test-Medium Tablet Fasted): A single 20-milligram (mg) LY2409021 tablet of a medium particle size administered orally, once in a fasted state, during Period 1, 2, or 3.
- LY2409021 Cohort 1 (Reference Capsules Fasted): A 20-mg LY2409021 dose administered orally, once in a fasted state, during Period 1, 2, or 3.
Arm/Group | LY2409021 Cohort 1 (Test-Medium Tablet Fasted) | LY2409021 Cohort 1 (Reference Capsules Fasted)
Number analyzed (Participants) | 16 | 15
nanograms*hour per milliliter (ng*hr/mL) | 65300 (20) | 62800 (38)
Statistical Analysis 1: Comparison: LY2409021 Cohort 1 (Test-Medium Tablet Fasted) vs LY2409021 Cohort 1 (Reference Capsules Fasted); Test type: Superiority or Other; Ratio of geometric least squares means = 1.03, 90% CI 2-sided [0.897 to 1.18] — AUC0-∞ was log-transformed and analyzed using a linear mixed effects model with fixed factors for formulation, sequence, and period, and random factor for participant

2. Primary Outcome: Pharmacokinetics, Maximum Concentration (Cmax): Medium Test Form to Reference Form
Time Frame: as for outcome 1
Population: Randomized participants in Cohort 1 who received the specified study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- LY2409021 Cohort 1 (Test-Medium Tablet Fasted): A single 20-mg LY2409021 tablet of a medium particle size administered orally, once in a fasted state, during Period 1, 2, or 3.
Arm/Group | LY2409021 Cohort 1 (Test-Medium Tablet Fasted) | LY2409021 Cohort 1 (Reference Capsules Fasted)
Number analyzed (Participants) | 16 | 15
nanograms per milliliter (ng/mL) | 779 (19) | 726 (41)
Statistical Analysis 1: Comparison: LY2409021 Cohort 1 (Test-Medium Tablet Fasted) vs LY2409021 Cohort 1 (Reference Capsules Fasted); Test type: Superiority or Other; Ratio of geometric least squares means = 1.06, 90% CI 2-sided [0.922 to 1.22] — Cmax was log-transformed and analyzed using a linear mixed effects model with fixed factors for formulation, sequence, and period, and random factor for participant

3. Secondary Outcome: Pharmacokinetics, Area Under the Concentration-Time Curve (AUC): Standardized High Fat Meal to Fasting
Description: AUC from time 0 to infinity (AUC0-∞).
Time Frame: as for outcome 1
Population: Randomized participants in Cohort 1 who received the specified study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*hr/mL)
Groups:
- LY2409021 Cohort 1 (Test-Medium Tablet Fed): A single 20-mg LY2409021 tablet of a medium particle size administered orally, once, immediately after a standardized high-fat meal, during Period 1, 2, or 3.
Arm/Group | LY2409021 Cohort 1 (Test-Medium Tablet Fed) | LY2409021 Cohort 1 (Test-Medium Tablet Fasted)
Number analyzed (Participants) | 18 | 16
nanograms*hour/milliliter (ng*hr/mL) | 67000 (18) | 65300 (20)
Statistical Analysis 1: Comparison: LY2409021 Cohort 1 (Test-Medium Tablet Fed) vs LY2409021 Cohort 1 (Test-Medium Tablet Fasted); Test type: Superiority or Other; Ratio of geometric least squares means = 1.02, 90% CI 2-sided [0.896 to 1.16] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Pharmacokinetics, Maximum Concentration (Cmax): Standardized High Fat Meal to Fasting
Time Frame: as for outcome 1
Population: Randomized participants in Cohort 1 who received the specified study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | LY2409021 Cohort 1 (Test-Medium Tablet Fed) | LY2409021 Cohort 1 (Test-Medium Tablet Fasted)
Number analyzed (Participants) | 18 | 16
nanograms per milliliter (ng/mL) | 785 (14) | 779 (19)
Statistical Analysis 1: Comparison: LY2409021 Cohort 1 (Test-Medium Tablet Fed) vs LY2409021 Cohort 1 (Test-Medium Tablet Fasted); Test type: Superiority or Other; Ratio of geometric least squares means = 1.01, 90% CI 2-sided [0.882 to 1.15] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Pharmacokinetics, Time to Maximum Concentration (Tmax)
Time Frame: as for outcome 1
Population: Randomized participants in Cohorts 1 and 2 who received the specified study drug.
Measure: Median (Full Range); unit: hour (hr)
Groups:
- LY2409021 Cohort 2 (Test-Low Tablet Fasted): A single 20-mg LY2409021 tablet of a low particle size administered orally, once in a fasted state, during Period 1, 2, or 3.
- LY2409021 Cohort 2 (Test-Medium Tablet Fasted): A single 20-mg LY2409021 tablet of a medium particle size administered orally, once in a fasted state, during Period 1, 2, or 3.
- LY2409021 Cohort 2 (Test-High Tablet Fasted): A single 20-mg LY2409021 tablet of a high particle size administered orally, once in a fasted state, during Period 1, 2, or 3.
Arm/Group | LY2409021 Cohort 1 (Reference Capsules Fasted) | LY2409021 Cohort 1 (Test-Medium Tablet Fed) | LY2409021 Cohort 1 (Test-Medium Tablet Fasted) | LY2409021 Cohort 2 (Test-Low Tablet Fasted) | LY2409021 Cohort 2 (Test-Medium Tablet Fasted) | LY2409021 Cohort 2 (Test-High Tablet Fasted)
Number analyzed (Participants) | 15 | 18 | 16 | 15 | 17 | 17
hour (hr) | 8.00 [4.00 to 12.00] | 8.00 [4.00 to 24.00] | 8.00 [4.00 to 12.00] | 4.00 [4.00 to 10.00] | 8.00 [4.00 to 18.00] | 8.00 [4.00 to 10.00]

6. Secondary Outcome: Pharmacokinetics, Area Under the Concentration-Time Curve (AUC): Low and High Particle Size to Medium Particle Size
Description: AUC from time 0 to infinity (AUC0-∞).
Time Frame: as for outcome 1
Population: Randomized participants in Cohort 2 who received the specified study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*hr/mL)
Arm/Group | LY2409021 Cohort 2 (Test-Low Tablet Fasted) | LY2409021 Cohort 2 (Test-High Tablet Fasted) | LY2409021 Cohort 2 (Test-Medium Tablet Fasted)
Number analyzed (Participants) | 15 | 17 | 17
nanograms*hour per milliliter (ng*hr/mL) | 73700 (16) | 69400 (18) | 73600 (17)
Statistical Analysis 1: Comparison: LY2409021 Cohort 2 (Test-Low Tablet Fasted) vs LY2409021 Cohort 2 (Test-Medium Tablet Fasted); Test type: Superiority or Other; Ratio of geometric least squares means = 0.993, 90% CI 2-sided [0.951 to 1.04] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: LY2409021 Cohort 2 (Test-High Tablet Fasted) vs LY2409021 Cohort 2 (Test-Medium Tablet Fasted); Test type: Superiority or Other; Ratio of geometric least squares means = 0.943, 90% CI 2-sided [0.905 to 0.983] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Pharmacokinetics, Concentration Maximum (Cmax): Low and High Particle Size to Medium Particle Size
Time Frame: as for outcome 1
Population: Randomized participants in Cohort 2 who received the specified study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | LY2409021 Cohort 2 (Test-Low Tablet Fasted) | LY2409021 Cohort 2 (Test-High Tablet Fasted) | LY2409021 Cohort 2 (Test-Medium Tablet Fasted)
Number analyzed (Participants) | 15 | 17 | 17
nanograms per milliliter (ng/mL) | 835 (20) | 793 (20) | 844 (20)
Statistical Analysis 1: Comparison: LY2409021 Cohort 2 (Test-Low Tablet Fasted) vs LY2409021 Cohort 2 (Test-Medium Tablet Fasted); Test type: Superiority or Other; Ratio of geometric least squares means = 0.980, 90% CI 2-sided [0.926 to 1.04] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: LY2409021 Cohort 2 (Test-High Tablet Fasted) vs LY2409021 Cohort 2 (Test-Medium Tablet Fasted); Test type: Superiority or Other; Ratio of geometric least squares means = 0.940, 90% CI 2-sided [0.891 to 0.993] — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Groups:
- LY2409021 Cohorts 1 and 2 (Test-Medium Tablet Fasted): A single 20-mg LY2409021 tablet of a medium particle size administered orally, once in a fasted state, during Period 1, 2, or 3.
Arm/Group | LY2409021 Cohort 1 (Reference Capsules Fasted) | LY2409021 Cohort 1 (Test-Medium Tablet Fed) | LY2409021 Cohort 2 (Test-Low Tablet Fasted) | LY2409021 Cohorts 1 and 2 (Test-Medium Tablet Fasted) | LY2409021 Cohort 2 (Test-High Tablet Fasted)
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/18 | 0/15 | 0/33 | 0/17
Other Adverse Events (participants affected / at risk) | 12/15 | 17/18 | 7/15 | 22/33 | 9/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2409021 Cohort 1 (Reference Capsules Fasted) (N=15) | LY2409021 Cohort 1 (Test-Medium Tablet Fed) (N=18) | LY2409021 Cohort 2 (Test-Low Tablet Fasted) (N=15) | LY2409021 Cohorts 1 and 2 (Test-Medium Tablet Fasted) (N=33) | LY2409021 Cohort 2 (Test-High Tablet Fasted) (N=17)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hunger (General disorders) | 1 (1) | 1 (2) | 3 (3) | 1 (1) | 2 (2)
Vessel puncture site haematoma (General disorders) | 4 (5) | 6 (10) | 2 (2) | 9 (12) | 3 (4)
Vessel puncture site pain (General disorders) | 2 (3) | 1 (1) | 0 (0) | 2 (3) | 2 (2)
Vessel puncture site reaction (General disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Vessel puncture site swelling (General disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Procedural site reaction (Injury, poisoning and procedural complications) | 6 (8) | 9 (13) | 3 (3) | 10 (15) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coagulation time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes